CLINICAL TRIAL: NCT04121975
Title: Concurrent Chemoradiotherapy Combined With Endostar for the Treatment of Locally Advanced Cervical Cancer, a Prospective, Single Arm Study
Brief Title: CCRT Combined With Endostar for the Treatment of Locally Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endo-CC-01
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; endostar protein; Endostatins; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemoradiotherapy (Experimental): Radiation:
  Radiotherapy was administered in 1.8-2.0 Gy fractions 5 times weekly to a total dose of 45-50 Gy.
  Drug: Endostar 30 mg/d was administered on days 1-5 every two weeks for 4 cycles.
  Drug: Cisplatin 30-40 mg/m2 was administered day 1, 8, 15, 22 and 29.
  Interventions: Radiation: Radiotherapy; Drug: Endostar; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy was administered in 1.8-2.0 Gy fractions 5 times weekly to a total dose of 45-50 Gy.
Drug: Endostar — 30 mg/d was administered on days 1-5 every two weeks for 4 cycles.
  Other Names: Recombinant human endostatin
Drug: Cisplatin — 30-40 mg/m2 was administered day 1, 8, 15, 22 and 29.

SUMMARY:
This was a prospective, single arm, phase 2 trial. Adult Patients with histologically confirmed locally advanced cervical cancer were enrolled to receive the treatment of concurrent chemoradiotherapy combined with Endostar. The primary endpoint was progression-free survival (PFS) rate at 1 year. The secondary endpoints were PFS, overall survival (OS) and safety.

DETAILED DESCRIPTION:
This was a prospective, single arm, phase 2 trial. Adult Patients with histologically confirmed locally advanced cervical cancer were enrolled to receive the treatment of concurrent chemoradiotherapy combined with Endostar. Radiotherapy was administered in 1.8-2.0 Gy fractions 5 times weekly to a total dose of 45-50 Gy. Endostar (30 mg/d) was administered on days 1-5 every two weeks for 4 cycles. Cisplatin (30-40 mg/m2) was administered day 1, 8, 15, 22 and 29. The primary endpoint was progression-free survival (PFS) rate at 1 year. The secondary endpoints were PFS, overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years old;
2. Histologically confirmed to be cervical squamous cell carcinoma;
3. Clinical stage IIB (need to have lymph node metastasis), IIIA, IIIB, IVA (2018 version of FIGO stage);
4. The ECOG PS score is 0 or 1;
5. At least one measurable (measured according to RECIST 1.1);
6. No distant organ metastasis confirmed by abdominal CT, chest CT, bone ECT, etc;
7. This treatment must be the first course of treatment;
8. The expected survival expectation is not less than 6 months;
9. The main organ function meets the following criteria within 7 days before treatment:

Blood routine examination standard (without blood transfusion within 14 days):

1. hemoglobin (HB) ≥ 90g / L;
2. neutrophil absolute value (ANC) ≥ 1.5 × 10 9 / L;
3. platelets (PLT) ≥ 80 × 10 9 / L.

Biochemical tests are subject to the following criteria:

1. total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
2. alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 times ULN;
3. serum creatinine (Cr) ≤ 1.5 times ULN or creatinine clearance (CCr) ≥ 60ml / min;

Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).

(10) Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy tests within 7 days prior to study enrollment And must be non-lactating patients; (11) Can understand the study and have signed an informed consent form;

Exclusion Criteria:

1. Patients with distant metastases;
2. Those suffering from other malignant tumors;
3. Have received cancer-related treatment such as radiotherapy or chemotherapy before enrollment;
4. Patients with contraindications to radiotherapy and chemotherapy, including serious infections or other complications such as severe cerebrovascular disease, mental illness and uncontrollable diabetes;
5. During pregnancy or lactation;
6. Those who have received targeted therapy;
7. Those who are in other drug trials;
8. Those with serious heart disease, including: congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina, myocardial infarction, severe heart valve disease, and refractory hypertension;
9. It is known that there is a hypersensitivity reaction to any component contained in the Endostar formulation;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) rate at 1 year | 1 year
  The rates of patients who were progression free at 1-year after enrollment

SECONDARY OUTCOMES:
Progression-free survival | 2 year
  Progression-free survival (PFS) is defined as the time from enrollment to disease progression or death from any cause.
Overall survival | 2 year
  Overall survival was defined as the time from enrollment to death from any cause
Treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  Treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hanmei Lou, PHD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China